CLINICAL TRIAL: NCT07313774
Title: A Randomized, Phase 3, Double-blind, Double-dummy, Active Comparator-controlled Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Linaprazan Glurate Compared to Lansoprazole in Maintenance of Healing in Participants With Healed Erosive Esophagitis (EE) Due to Gastroesophageal Reflux Disease (GERD) of Los Angeles (LA) Grades A to D
Brief Title: A Study Comparing the Effect and Safety of Linaprazan Glurate to Lansoprazole in Maintenance of Healing in Participants With Healed Erosive Esophagitis (EE) Due to Gastroesophageal Reflux Disease (GERD)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CX842A2303; 2025-522750-39-00 (EU CTIS Number); U1111-1324-0039 (Other: World Health Organization)
Record Dates: First submitted 2025-12-19; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Linaprazan glurate - High dose (Experimental)
  Interventions: Drug: Linaprazan glurate - High dose
- Linaprazan glurate - Low dose (Experimental)
  Interventions: Drug: Linaprazan glurate - Low dose
- Lansoprazole (Active Comparator)
  Interventions: Drug: Lansoprazole - Marketed approved dose

INTERVENTIONS:
Drug: Linaprazan glurate - High dose — Linaprazan glurate - High dose administered as per protocol
  Arms: Linaprazan glurate - High dose
Drug: Linaprazan glurate - Low dose — Linaprazan glurate - Low dose administered as per protocol
  Arms: Linaprazan glurate - Low dose
Drug: Lansoprazole - Marketed approved dose — Lansoprazole administered as per protocol
  Arms: Lansoprazole

SUMMARY:
The goal of this clinical trial is to investigate how well linaprazan glurate can maintain healed erosive esophagitis (EE) caused by GERD in participants who have participated in a prior healing trial, compared to lansoprazole (an approved treatment for GERD). Researchers will also examine:

* the effect of linaprazan glurate on heartburn symptoms compared to lansoprazole.
* whether linaprazan glurate treatment is safe and tolerable, based on symptoms and procedures such as blood and urine tests, endoscopy, and electrocardiograms (measure the heart's electrical activity). Endoscopy means that the doctor will insert a thin, flexible tube with a camera down the throat to look at each participant's esophagus area and collect small tissue samples (called biopsies).
* the side effects that may happen during treatment with linaprazan glurate.

Participants must be between 18 to 80 years old and have participated in a prior healing trial with healed EE (due to GERD) confirmed by an endoscopy either from the prior healing trial or from the initial period of this trial. Participants cannot participate if they are not healed, had to stop trial treatment because of a side effect in a prior healing trial, or if they have a condition that could make it unsafe.

The study is a randomized, double-blind, active comparator-controlled clinical trial lasting for almost 14 months. Randomized means that participants are assigned by chance (like flipping a coin) to one of the treatment groups and double-blind means neither the participants nor the study team will know which treatment is given. Participants will be placed into one of three groups:

* Linaprazan glurate - High dose
* Linaparazan glurate - Low dose, and
* Lansoprazole - marketed approved dose Everyone will take a total of 2 tablets and 1 capsule orally every day for up to 52 weeks. The tablets and capsule will be separated into a morning dose and an evening dose. Some tablets or capsules will be placebos (look like medicine but contain no active drug).

Participants will complete several questionnaires on an electronic device during treatment. An endoscopy will be performed after 24 weeks of treatment to determine if healing has been maintained. If healing has been maintained, the participant will continue taking trial treatment and another endoscopy will be performed at 52 weeks. If healing has not been maintained at 24 weeks or if the participant has reached 52 weeks, the participant will stop taking trial treatment and return for a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

An individual who has participated in a preceding linaprazan glurate healing trial will be asked to participate in this maintenance trial if the following criteria apply:

1. The participant understands and voluntarily signs an Informed Consent Form (ICF) prior to initiation of any trial-related assessments/procedures.
2. The participant has a healed EE as assessed by central review of endoscopic examination either from the last regular visit in a preceding phase 3 healing trial OR from the Run-in Period to the present maintenance trial.
3. The participant is willing and able to comply with all aspects of the protocol (including endoscopies, tablet and capsule swallowing, electronic device [e-device] completion, etc.).

Exclusion Criteria:

An individual who has participated in a preceding linaprazan glurate phase 3 healing trial can be enrolled in this maintenance trial unless they meet any of the following exclusion criteria:

1. EE as graded from the endoscopy during the Run-in Period (only applicable for participants with previous endoscopy >14 days before the last regular visit in the preceding healing trial).
2. Solitary esophageal ulcer in the proximal two-thirds of the esophagus, untreated Barrett's esophagus or any other condition affecting the esophagus, including eosinophilic esophagitis; esophageal varices; viral or fungal infection; esophageal stricture.*

   *Note: Participants with diagnosis of Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) are eligible to participate, unless history of dilatation within 3 months of the Run-in Period.
3. Significant noncompliance with protocol-specified procedures or treatment in the preceding healing trial as judged by the Investigator.
4. Adverse event (AE) resulting in premature discontinuation of IP in the preceding healing trial.
5. History or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, neurological disease or disorder, or psychiatric diagnosis which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the trial results or the participant's ability to participate in the trial. The following examples are conditions that would exclude the participant from participating:

   1. History of myocardial infarction/ acute coronary syndrome within 3 months prior to the M0 visit.
   2. History of ventricular arrhythmia or implanted cardioverter defibrillator
   3. Symptomatic congestive heart failure (New York Heart Association [NYHA] class 3-4)
   4. Family history of/ diagnosis of hereditary arrhythmia syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Maintained healing of EE after 24 weeks as assessed by central reading of endoscopy. | From enrollment to the end of 24 weeks of treatment

IPD SHARING:
Plan to Share IPD: No